CLINICAL TRIAL: NCT03049579
Title: Immune System Stimulation by Probiotic Food Supplementation: a Double-blind, Randomized, Controlled, Parallel-designed, Prospective Trial
Brief Title: Immune System Stimulation by Probiotic Food Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Wei Chuan Foods Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-SC-09-WQ-002
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Flu Symptom
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weiquan Yogurt with probiotics (Experimental): Weiquan Yogurt with probiotics contained Lactobacillus paracasei (108 colony forming units (CFU)/ml), Lactobacillus casei 431® (108 CFU/ml) and Lactobacillus fermentum PCC® (106 CFU/ml)
  Interventions: Dietary Supplement: Weiquan Yogurt with probiotics
- Weiquan Yogurt without probiotics (Placebo Comparator): Weiquan Yogurt devoid of probiotics, but otherwise similar to the experimental product.
  Interventions: Dietary Supplement: Weiquan Yogurt without probiotics

INTERVENTIONS:
Dietary Supplement: Weiquan Yogurt with probiotics — 150 ml daily consumption for a total of 12 weeks
  Arms: Weiquan Yogurt with probiotics
Dietary Supplement: Weiquan Yogurt without probiotics — 150 ml daily consumption for a total of 12 weeks
  Arms: Weiquan Yogurt without probiotics

SUMMARY:
The purpose of this study is to investigate the effects of a probiotic supplementation on adult volunteers with having caught the common cold more than 4 times in the past year. This study is a single center, double-blind, randomized, controlled, parallel-designed, prospective trial. Subjects received a probiotic drink containing probiotics of Lactobacillus paracasei (108 colony forming units (CFU)/ml), Lactobacilluscasei431® (108CFU/ml) and Lactobacillus fermentiumPCC® (106CFU/ml) or an identical placebo without probiotics for a 12-week study period.

The incidence of flue and cold during the study period were compared between study groups.

Blood and fecal samples were collected at baseline and at the end of the intervention. Fecal samples were collected for the secretory immunoglobulin A (sIgA) analysis. Blood sample was drawn for interferon γ (IFN-γ), interleukin 4 (IL-4), interleukin 10 (IL-10), immunoglobulin A (IgA), immunoglobulin G (IgG) and immunoglobulin M (IgM) analysis.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 25 to 45 years old;
* having caught the common cold or flu at least 4 to 6 times in the past calendar year;
* signed the informed consent forms before entering the study;
* fully understood the risks and potential benefits in participating this study.

Exclusion Criteria:

* were diagnosed with the decreased immunity caused by any diagnosed chronic illness;
* having any gastrointestinal illness with medical treatment at the time of being enrolled;
* having any diagnosed respiratory illness with similar symptoms as the common cold and flu;
* currently taking any pain killer drug;
* having received any vaccine for the upper respiratory infection within 6 months before enrollment;
* having received any purgative drug or digestion related drug within 2 weeks before enrollment;
* having taken any dairy product containing prebiotics and probiotics within 10 days before enrollment;
* currently taking any preventive drug for upper respiratory infection;
* having received any drug which has impact with the immune system such as antibiotics within 3 months before enrollment;
* alcoholic or addicted to any drug;
* pregnant or breastfeeding mothers;
* having participated another clinical trial within 3 months before enrollment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Incidence of flue symptoms during the study | end of week 12
  Body temperature≥38.0℃, and have one or more symptoms of cough, runny nose, throat pain, headache, muscle pain, weak feeling, hard to breath, chest pain or loss of appetite.

SECONDARY OUTCOMES:
Incidence of cold symptoms during the study | end of week 12
  Body temperature<38.0℃, and have one or more symptoms of cough, runny nose, throat pain, headache, muscle pain, weak feeling, hard to breath, chest pain or loss of appetite.
Number of accumulated days of having cold symptoms during the study | End of week 12
  The total number of days of having one or more symptoms of cough, runny nose, throat pain, headache, muscle pain, weak feeling, hard to breath, chest pain or loss of appetite during the 12 week study period.
Serum IFN-γ concentration | Baseline, end of week 12
  Interferon gamma (unit: pg/ml)
Serum IL-4 concentration | Baseline, end of week 12
  Interleukin 4 (unit: ng/ml)
Serum IL-10 concentration | Baseline, end of week 12
  Interleukin 10 (unit: pg/ml)
Serum IgA concentration | Baseline, end of week 12
  Immunoglobulin A (unit: g/L)
Serum IgG concentration | Baseline, end of week 12
  Immunoglobulin G (unit: g/L)
Serum IgM concentration | Baseline, end of week 12
  Immunoglobulin M (unit: g/L)
Fecal sIgA concentration | Baseline, end of week 12
  Secretory Immunoglobulin A (unit: ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Director — Sprim (Shanghai) Consulting Co., Ltd.

IPD SHARING:
Plan to Share IPD: No